CLINICAL TRIAL: NCT01506206
Title: ON/OFF Stimulation and Impulsivity in Patients With Deep Brain Stimulators
Status: Withdrawn | Type: Observational
Why Stopped: Study was not funded and never enrolled participants.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Darin Dougherty, MD, Associate Professor of Psychiatry, Massachusetts General Hospital
Other Study IDs: 2011P002546
Record Dates: First submitted 2012-01-05; First posted 2012-01-09 (Estimated); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Obsessive Compulsive Disorder; Major Depressive Disorder
Keywords: Deep Brain Stimulation; Impulsivity
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Depressive Disorder, Major; Impulsive Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with Deep Brain Stimulators: Patients with deep brain stimulation for either major depressive disorder (MDD) or obsessive compulsive disorder (OCD).
- Patients with MDD or OCD: Patients with MDD or OCD who do not have a deep brain stimulator.

SUMMARY:
The investigators propose a test of causality by examining a cohort of patients undergoing deep brain stimulation (DBS) within the ventral striatum. The investigators will examine behavior on and off stimulation across a range of tasks that index different forms of impulsivity. Patients will be studied in both the ON and OFF state - that is, they will be tested during active deep brain stimulation and 30 min to 1 hour after stimulation has been stopped (order of state will be counterbalanced across subjects). The investigators specific aim is to test the hypothesis that enhancing ventral striatal signaling (i.e. ON-state DBS) will cause more impulsive patterns of behavior across several impulsivity tasks. The investigators predict that ventral striatal DBS will increase stop-signal reaction time on the stop-signal task and commission errors on the Go/NoGo task, and increase delay aversion in a delay discounting paradigm.

DETAILED DESCRIPTION:
The study will take place at a clinical office in the Charlestown Navy Yard (CNY), and will consist of 4 or 4.5 hour visit. Study staff will schedule a convenient time for patients to arrive, or the research visit may be paired with a regularly scheduled DBS programming visit. A member of the Division of Neurotherapeutics authorized to manipulate DBS programming will turn the device ON and OFF during the study. The subject's therapeutic parameters of the DBS system will not be changed. The subject will be asked to complete 2 questionnaires. Following these questionnaires, DBS stimulation will be turned off and a member of the study staff will teach the subjects to perform the following tasks on the computer:

Stop-Signal Task To measure "impulsive action," the investigators will use the stop-signal task (SST), a well-validated measure of response inhibition known to be impaired in substance abusers. In each of the 192 trials (3 blocks of 64; 10s interval between blocks, 2s ISI), subjects see a fixation cue (250ms) that is replaced by a shape (square or circle). Participants are told to make a shape judgment by pressing the appropriate computer key. On no-signal trials (75%), subjects are instructed to respond to the stimulus as fast and accurately as possible. On stop-signal trials (25%), the stimulus is followed by an auditory stop signal, and subjects are instructed to withhold responding. On stop-signal trials, a stop signal is presented after a variable delay (SSD), initially set at 250 msec and adjusted continuously with a staircase procedure by 50ms depending on whether inhibition is successful (increases) or unsuccessful (decreases). The paradigm will be administered using precompiled software provided by Gordon Logan, which automatically analyzes all relevant dependent variables (e.g stop-signal reaction time [SSRT] and GoRT). This task takes approximately 20 minutes.

Rewarded Variant This task is a variant of the above, with an inclusion of a "points possible cue" (2 or 50 points) for 500 ms, and followed by a brief delay (500-1500 ms) prior to the target. The task will be presented in 13 blocks. The first contains only go trials, from which the initial SSD will be calculated. The 12 subsequent blocks each consist of 40 trials; 18 standard go trials, 12 high reward (HR) go trials, 6 standard stop trials, and 4 HR stop trials, presented in random order. The SSD will be determined by a simple staircase-tracking algorithm as described by Logan, in which the SSD is adjusted up or down by 25 ms in order to establish an SSD that produces 50% accuracy of successful performance, with separate staircases calculated for the HR and standard trials. Outcome measures are the standard and high reward GoRTs, the standard and HR SSRTs, and the proportion of responses that would have been unsuccessfully stopped on HR trials if the standard SSD were utilized instead of the HR SSD.

Rewarded Go/NoGo Task In this task, participants are asked to make, or withhold, a button press to one of six stimuli (shapes), that correspond to six trial types: Go (no reward), Go (low reward), Go (high reward), NoGo (no reward), NoGo (low reward), NoGo (high reward). Participants are asked to press a button for Go stimuli and withhold a button press for NoGo stimuli. The ratio of Go stimuli to NoGo stimuli is approximately 15:1. Participants win money for correctly pressing a button for Go stimuli and for withholding a response for NoGo stimuli; conversely, they lose money for failing to respond to a Go stimuli or for failing to withhold a response to NoGo stimuli. There are 1260 trials, and each lasts 1 second. The task takes about 20 minutes to complete. Task may be administered without reward contingencies. In this case, there will only be two trial types: Go and NoGo.

Delay Discounting Task To measure "impulsive choice" the investigators will use a delay-discounting (DD) paradigm101. On each trial, participants make a binary choice between a smaller/sooner and a larger/later reward. The delay of the sooner reward is set as today, 2 weeks, & 1 month; the delay of the later reward ranges from 2 to 6 weeks after the early reward. The sooner reward is from 1% to 50% less than the late reward (max = $40). Participants will complete approximately 80 trials. Participants are told that two of their choices will be randomly selected for payout at the appropriate time. Outcome variables include the proportion of choices for immediate/sooner rewards, as well as discounting parameter k, obtained by fitting choice data for each subject to a hyperbolic discount function. The task takes approximately 15 minutes to complete.

30 minutes after turning OFF DBS stimulation, participants will either remain in the OFF condition or will have the DBS turned ON, depending on their counter-balanced condition assignment. Subjects will complete the tasks above in the first condition. Following task completion, subjects will have DBS stimulation turned OFF or ON (again, depending on condition assignment). After 30 minutes, participants will complete the same tasks in the second condition. Following retesting, participants that were in the OFF condition will return to ON DBS stimulation.

The investigators will be using the implanted pulse generator to deliver a safe current. Because the investigators are not changing the therapeutic parameters of stimulation, subjects should not experience any changes during the ON condition. Should any discomfort arise in the OFF condition, the subject will be able to terminate the study and return to the ON condition immediately. The computer will register the subject's performance.

Electroencephalography recordings (EEG) will be acquired during performance of the aforementioned tasks. Continuous EEG data will be sampled at a maximum of 1024Hz using a 64-electrode cap. Eye movement artifacts will be assessed using bipolar electrodes.

Patients with just major depressive disorder or obsessive compulsive disorder will also be recruited as a control group for the patients with deep brain stimulation.

ELIGIBILITY:
DBS Patients:

Inclusion Criteria:

* Deep brain stimulator implantation performed at least three months prior to study

Exclusion Criteria:

* Subjects unable to visualize stimulus objects with correction
* Dementia or other known cognitive deficit

Psychiatric Patients:

Inclusion Criteria:

* Right-handed (as determined by the Handedness Inventory; Oldfield, 1971)
* Normal or corrected-to normal vision and hearing
* Current diagnosis of MDD or OCD

Exclusion Criteria for Patients:

* Clinical history of bipolar disorder
* Current or past psychotic disorder
* Gross structural brain damage
* Cognitive impairment that would affect a participant's ability to give informed consent
* Current substance abuse, or abuse within the past 3 months
* Clinical history of severe personality disorder
* Imminent risk of suicide or an inability to control suicide attempts
* Evidence of dementia or other significant cognitive impairment on neuropsychological evaluation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Deep Brain Stimulators Patients with Major Depressive Disorder or Obsessive-Compulsive Disorder and no DBS
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-02; Primary Completion 2024-01-10 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Impulsive Action | 2 hours
  As measured by the Go/No Go task

SECONDARY OUTCOMES:
Impulsive Choice | 2 hours
  As measured by delayed discounting task

CONTACTS AND LOCATIONS:
Overall Officials: Darin D Dougherty, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Massachusetts General Hospital, Charlestown, Massachusetts